CLINICAL TRIAL: NCT02045771
Title: A Pragmatic Randomized Trial to Investigate the Effectiveness of BehaviouRal ActiVation Group Therapy in Reducing dEpressive Symptoms and Improving Quality of Life in Patients With Depression: BRAVE Pilot Study
Brief Title: A Pilot Study to Assess the Effectiveness of BehaviouRal ActiVation Group Program in Patients With dEpression: BRAVE
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Zainab Samaan (Zena), Assistant Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVE Pilot Trial
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2017-01

CONDITIONS: Depression
Keywords: Depression; Behavioral Activation
MeSH Terms: conditions — Depression | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Support Group (Control Group) (Other): In addition to usual care, the control group will be offered a support group therapy format delivered at the same place, same visit frequency and duration of program as the intervention group. This support group is intended to simulate the intervention group format to minimize risk of biased estimate of BA effectiveness by reducing the potential placebo effect which can be seen due to frequent clinic visits and having additional attention beyond usual care.
  Interventions: Behavioral: Support Group
- Behavioral Activation (Experimental): Originally a component of cognitive therapy, behavioural activation is the use of strategies such as activity scheduling, master/pleasure ratings, and graded task assignments to change one's perception of specific situations. It involves the use of activities to improve life situations or depressed mood.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral activation is a therapy, which has been shown to be quite effective in the treatment of depression (Kanter, Manos et al. 2010; Martell, Dimidjian et al. 2010). Although previous therapies have focused more on the cognitive element, behavioural activation on its own has also been significantly effective for depression treatment (Jacobson, Dobson et al. 1996). The treatment works by increasing behaviours that help a patient with depression interact with an environment and providing consequences to positively reinforce "antidepressant behaviour" (Martell, Dimidjian et al. 2010).
  Arms: Behavioral Activation
Behavioral: Support Group — In addition to usual care, the control group will be offered a support group therapy format delivered at the same place, same visit frequency and duration of program as the intervention group. This support group is intended to simulate the intervention group format to minimize risk of biased estimate of BA effectiveness by reducing the potential placebo effect which can be seen due to frequent clinic visits and having additional attention beyond usual care.
  Arms: Support Group (Control Group)

SUMMARY:
The study's primary goal is to assess the effectiveness of behavioural activation in reducing depressive symptoms and re-integrate patients with depression into their personal and professional lives thus improving quality of life and helping in attaining and maintaining remission of depression. It is aimed at helping patients re-engage with several life areas that they may have lost in the course of depressive illness. The intervention is centred on behavioural activation (BA) with complementary interventions including recreation activities, and behavioural modifications. The study question is: in patients with depressive disorder attending a specialized hospital based mood disorders clinic, does the addition of behavioural activation program delivered in a group format improve depressive symptoms and quality of life compared to treatment as usual after 18 weeks of treatment? Study investigators hypothesize that behavioural activation is an effective treatment for depressive disorder in patients with depression.

DETAILED DESCRIPTION:
This is a pilot study, a mixed-methods design including an open label pragmatic randomized trial and a qualitative grounded theory approach. Participants will be randomized to Behavioural Activation (BA) (intervention) or support group (control) in addition to treatment as usual. The qualitative component will be used to gather participant's experiences, beliefs and opinions about two topics: 1) the experience of participating in the behavioural activation program and 2) their evolving perceptions of their individual depressive illness and quality of life. Based on the analysis of qualitative data pertaining to the first topic, the behavioural activation program may be modified for the main trial, to respond to patient needs and feedback, in the spirit of delivering truly patient centered care. The qualitative study will involve multiple interviews and focus groups which will take place before, during, and after the pilot intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder
* Must be able to provide written informed consent
* Must be able to attend program sessions

Exclusion Criteria:

* Inability to understand written and spoken English
* Primary diagnosis other than Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rates, data completion, and resource utilization. | Baseline, Week 18
  Assess feasibility of the study process in terms of recruitment, retention, number of sessions completed, average group size and data completion.

SECONDARY OUTCOMES:
Qualitative study feedback. | At weeks 2 and 10 of the 18 week program.
  The qualitative component of the pilot study is to assess the need to modify the protocol for the main trial based on participant's feedback.
Feasibility of economic evaluation using the EuroQol economic evaluation tool; EQ-5D-5L. | Baseline, Week 18
  EQ-5D-5L is a commonly used standardized generic measure of health and economic appraisal in a variety of clinical conditions. This will assist in the exploration of economic evaluation of the behavioral activation program in the main trial. the EQ-5D-5L consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The response to each dimension is a five-level severity ranging from "no problem" to "extreme problem".

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Samaan, MBChB PhD MRCPsych, Principal Investigator — McMaster University and St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Wampold BE, Minami T, Tierney SC, Baskin TW, Bhati KS. The placebo is powerful: estimating placebo effects in medicine and psychotherapy from randomized clinical trials. J Clin Psychol. 2005 Jul;61(7):835-54. doi: 10.1002/jclp.20129. PMID 15827993
- [Derived] D'Elia A, Bawor M, Dennis BB, Bhatt M, Litke K, McCabe K, Whattam J, Garrick L, O'Neill L, Simons S, Chalmers S, Key B, Goyert S, Laplante P, Vanstone M, Xie F, Guyatt G, Thabane L, Samaan Z. Feasibility of behavioral activation group therapy in reducing depressive symptoms and improving quality of life in patients with depression: the BRAVE pilot trial. Pilot Feasibility Stud. 2020 May 7;6:61. doi: 10.1186/s40814-020-00596-z. eCollection 2020. PMID 32411381
- [Derived] Chum J, Kim MS, Zielinski L, Bhatt M, Chung D, Yeung S, Litke K, McCabe K, Whattam J, Garrick L, O'Neill L, Goyert S, Merrifield C, Patel Y, Samaan Z. Acceptability of the Fitbit in behavioural activation therapy for depression: a qualitative study. Evid Based Ment Health. 2017 Nov;20(4):128-133. doi: 10.1136/eb-2017-102763. Epub 2017 Oct 22. PMID 29056608
- [Derived] Samaan Z, Dennis BB, Kalbfleisch L, Bami H, Zielinski L, Bawor M, Litke K, McCabe K, Whattam J, Garrick L, O'Neill L, Tabak TA, Simons S, Chalmers S, Key B, Vanstone M, Xie F, Guyatt G, Thabane L. Behavioral activation group therapy for reducing depressive symptoms and improving quality of life: a feasibility study. Pilot Feasibility Stud. 2016 Apr 29;2:22. doi: 10.1186/s40814-016-0064-0. eCollection 2016. PMID 27965841
- [Derived] Samaan Z, Litke K, McCabe K, Dennis B, Whattam J, Garrick L, O'Neill L, Tabak TA, Simons S, Chalmers S, Key B, Vanstone M, Xie F, Guyatt G, Thabane L. A pragmatic pilot randomized trial to investigate the effectiveness of behavioural activation group therapy in reducing depressive symptoms and improving quality of life in patients with depression: the BRAVE pilot trial protocol. Pilot Feasibility Stud. 2015 Nov 10;1:39. doi: 10.1186/s40814-015-0034-y. eCollection 2015. PMID 27965817